CLINICAL TRIAL: NCT00005901
Title: A Trial of Pamidronate in Children With Osteogenesis Imperfecta
Brief Title: Pamidronate to Treat Osteogenesis Imperfecta in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000136; 00-CH-0136 (Other: NIH NICHD IRB)
Record Dates: First submitted 2000-06-06; First posted 2000-06-07 (Estimated); Results first posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Osteogenesis Imperfecta
Keywords: Bisphosphonates; Growth Hormone; Bone Density; Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta | interventions — Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pamidronate every 3 months for 3 years (Active Comparator): Subjects who received Pamidronate every 3 months for 3 years.
  Interventions: Drug: Pamidronate (Aredia)
- Pamidronate every 6 months for 3 years (Active Comparator): Subjects who received Pamidronate every 6 months for 3 years.
  Interventions: Drug: Pamidronate (Aredia)

INTERVENTIONS:
Drug: Pamidronate (Aredia) — Patients receive a dose of 1mg/kg/cycle (3-day infusion = 1 cycle)

SUMMARY:
This study will evaluate the effect of pamidronate a drug that decreases bone resorption (breakdown) on osteogenesis imperfecta. This is a genetic disorder of collagen, the major protein in bone. The abnormal collagen causes weak bones, and children with severe osteogenesis imperfecta sustain many fractures throughout their lives. They also have growth deficiency, curvature of the spine, crumbling teeth, hearing loss, easy bruising and heart and lung problems. The study will compare bone density, quality and strength, final adult height, trunk height, and functional ability in children who receive 1) pamidronate every 3 months, 2) pamidronate every 3 months + growth hormone injections, 3) pamidronate every 6 months, or 4) pamidronate every 6 months + growth hormone injections.

Children 2 years of age and older with severe osteogenesis imperfecta (types III and IV) may be eligible for this study. Those enrolled will be randomly assigned to groups according to age; children two to four years of age will be randomly assigned to receive pamidronate every 3 or every 6 months. Children four years of age and older may participate in the growth hormone treatment groups. These children will continue on growth hormone until they reach their adult height or fail to grow as much as would be expected for someone on growth hormone.

Patients will be followed in the clinic every 3 months for a history, physical examination, X-rays, blood tests, and measurements (weight, head circumference, and bone lengths). Children will receive a 3 to 4 hour infusion of pamidronate through an intravenous catheter (thin flexible tube placed in a vein) once a day for 3 days each visit. (Once inserted, the catheter is left in place to avoid multiple needle sticks for administering the drug and collecting blood samples.) Children who are taking growth hormone will be given the drug at the first treatment visit. At that time, the accompanying parent will be instructed on how to mix the drug and give injections. The child receives an injection 6 days a week (Sunday off).

DETAILED DESCRIPTION:
Osteogenesis imperfecta is an inherited disorder of connective tissue in which affected individuals synthesize abnormal type I collagen. This results in the formation of abnormal bone matrix and a predisposition to bony fractures. Many unsuccessful attempts have been made to increase the bone mineral density of these individuals in the hope that this will improve the strength of their bones and result in a decreased fracture rate.

Bisphosphonates are synthetic analogs of pyrophosphate which have an affinity for hydroxyapatite. These drugs act primarily on osteoclasts, impairing the development of immature osteoclasts and the function of mature osteoclasts, as well as depressing chemical signaling to adjacent cells, resulting in a shift in the balance of deposition and resorption in bone. Conditions for which bisphosphonates are being used in children include four broad categories, 1) a primary defect in bone mineralization 2) bone matrix abnormalities 3) bone abnormalities due to systemic disease or the effects of treatment of systemic disease or 4) significant soft tissue calcification with no bone abnormality.

Pamidronate, an aminobisphosphonate, is a potent inhibitor of bone resorption. The purpose of this protocol is to evaluate the effectiveness of pamidronate in children with types III and IV osteogenesis imperfecta when the cycle time is varied. We plan to compare children treated with pamidronate on an every-three-month infusion cycle to children treated every six months with the same dose per infusion. We also plan to continue to compare children treated with pamidronate and growth hormone to children treated with pamidronate alone.

ELIGIBILITY:
INCLUSION CRITERIA:

Children enrolled in this study will be limited to those with Sillence types III and IV OI, as determined by clinical and genetic criteria.

Most of the children who will be included in this study are already enrolled in the protocols Evaluation and Intervention for Ambulation, Growth, and Basilar Invagination in Osteogenesis Imperfecta (97-CH-0064) and Growth Hormone Therapy in Osteogenesis Imperfecta (92-CH-0034).

Screening of candidates will be based on telephone interviews with a parent, and referral records to include: AP and lateral radiographs of the lower extremities and spine, and family, developmental, fracture and medical history. An NIH clinical screening evaluation will be performed for those children who appear to have a history consistent with OI under protocol 04-CH-0077, Screening of and Diagnosis of Patients with Connective Tissue Disorder . Patients admitted for this screening visit who are less than four years of age as well as those older than 4 years of age but not meeting the criteria for inclusion in the growth hormone protocol, protocol 92-CH-0034, will be considered for enrollment in protocol 97-CH-0064 (Evaluation and Intervention for Ambulation, Growth and Basilar Invagination in OI), those older than four years who meet the criteria will be considered for co-enrollment in protocol 92-CH-0034.

The inclusion criteria for protocol 92-CH-0034 are as follows: patients must have a clinical/biochemical diagnosis of osteogenesis imperfecta types III or IV, height less than third percentile for age, and radiological evidence that long bone epiphyses have not yet fused.

Patients are excluded from protocol 92-CH-0034 if they have scoliosis of greater than 40 degrees unless scoliosis has been stable over the past two years, or evidence of severe basilar invagination.

Patients with previous exposure to bisphosphonates in outside trials will be considered for participation in this trial.

EXCLUSION CRITERIA:

Inability to comply with the visit schedule, maintenance of the physical therapy program, and ability to administer and comply with GH injections are central to our analysis of the outcomes of this study. Failure to comply with these conditions will constitute exclusion criteria.

Pregnancy.

Patients that have had or will have surgery to place instrumentation in the spine (i.e. result of spine fusion).

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2000-06; Primary Completion 2014-05 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan C Marini, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Marini JC. Osteogenesis imperfecta: comprehensive management. Adv Pediatr. 1988;35:391-426. No abstract available. PMID 3055864
- [Background] Prockop DJ, Kivirikko KI. Heritable diseases of collagen. N Engl J Med. 1984 Aug 9;311(6):376-86. doi: 10.1056/NEJM198408093110606. No abstract available. PMID 6146097
- [Background] Marini JC, Bordenick S, Heavner G, Rose S, Chrousos GP. Evaluation of growth hormone axis and responsiveness to growth stimulation of short children with osteogenesis imperfecta. Am J Med Genet. 1993 Jan 15;45(2):261-4. doi: 10.1002/ajmg.1320450223. PMID 8456815
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-CH-0136.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Comparator: 1: Receives treatment every 3 months
- Active Comparator: 2: Receives treatment every 6 months.
Period: Overall Study
Arm/Group | Active Comparator: 1 | Active Comparator: 2
Started | 19 | 15
Completed | 19 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Comparator: 1: Subjects who received Pamidronate every 3 months for 3 years.
- Active Comparator: 2: Subjects who received Pamidronate every 6 months for 3 years.
- Total: Total of all reporting groups
Arm/Group | Active Comparator: 1 | Active Comparator: 2 | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19 | 15 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 11 | 6 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 16 | 14 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 14 | 13 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5
Bone Mineral Density in Response to Pamidronate [Mean (Standard Deviation); unit: Z-score] — Dual-energy X-ray Absorptiometry (DXA) measurements were obtained using a Hologic QDR 4500 densitometer and low density software package. Measurements have a precision of 0.011 SD. Raw measurements were converted to Z-scores for analysis using the manufacturer's reference standards for age and pubertal status.
  Z-score | -5.01 (1.79) | -5.68 (0.96) | -5.32 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: Dual-energy X-ray Absorptiometry (DXA) measurements were obtained using a Hologic QDR 4500 densitometer and low density software package. Measurements have a precision of 0.011 SD. Raw measurements were converted to Z-scores for analysis using the manufacturer's reference standards for age and pubertal status.
Time Frame: Baseline vs. 12 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -3.54 (1.51) | -4.98 (1.16)

2. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: as for outcome 1
Time Frame: Baseline vs. 18 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -3.71 (1.4) | -4.65 (1.06)

3. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: as for outcome 1
Time Frame: Baseline vs. 24 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -3.48 (1.31) | -4.7 (1.37)

4. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: as for outcome 1
Time Frame: Baseline vs. 30 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -3.48 (1.09) | -4.05 (1.28)

5. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: as for outcome 1
Time Frame: Baseline vs. 36 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -3.31 (1.22) | -4.18 (1.67)

6. Primary Outcome: Change in Bone Mineral Density in Response to Pamidronate
Description: as for outcome 1
Time Frame: Baseline vs. 6 months after first dose
Population: All subjects received Pamidronate for 3 years.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Pamidronate Every 3 Months for 3 Years | Pamidronate Every 6 Months for 3 Years
Number analyzed (Participants) | 19 | 15
Z-score | -4.01 (1.79) | -4.98 (1.15)

ADVERSE EVENTS:
Time Frame: 3 years.
Arm/Group | Active Comparator: 1 | Active Comparator: 2
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Comparator: 1 (N=19) | Active Comparator: 2 (N=15)
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No